CLINICAL TRIAL: NCT02951091
Title: The Master Protocol for Biomarker-Integrated Umbrella Trial in Advanced Gastric Cancer
Brief Title: Biomarker-Integrated Umbrella, Advanced Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Sun Young Rha, professor, Yonsei University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2015-0616
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2024-12-30 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Biomarker-integrated multi-arm with shared standard of care (SOC) control arm
Oversight: Data Monitoring Committee: No

ARMS (2):
- biomarker group (Experimental): 400 Her-2 (-) metastatic/recurrent gastric cancer patients will be centrally screened for druggable targets [Epstein-Barr virus, Microsatellite instability, HER2, EGFR, c-MET, and PTEN] by immunohistochemistry and in situ hybridization during first line chemotherapy. At the time of second line treatment, patients will be randomized to the biomarker vs control group as 4: 1 ratio. The biomarker group will be offered for entry into a specific protocol based on their molecular cohort and treated with specific targeted agents in combination with weekly paclitaxel; 1) EGFR cohort (EGFR 2+ or EGFR 3+) for pan-ERBB inhibitor (afatinib), 2)PTEN loss cohort (PTEN score less than 100) for PIK3CB inhibitor (GSK2636771), 3) PD-L1 positive, MSI-high, or EBV positive cases for nivolumab, 4) none for weekly paclitaxel.
  Interventions: Other: biomarker screening
- control group (Active Comparator): Patients will be randomized to the biomarker vs control group (standard of care; paclitaxel) as 4:1 ratio.
  Interventions: Other: biomarker screening

INTERVENTIONS:
Other: biomarker screening — immunohistochemistry and in situ hybridization

SUMMARY:
In-depth understanding of molecular characteristics of gastric cancer enabled us to realize personalized medicine with targeted agents in gastric cancer treatment.

The investigators initiated open-label, randomized, controlled phase II, multi-arm trial comparing targeted therapy based on tumor molecular profiling with standard paclitaxel therapy as second line treatment.

DETAILED DESCRIPTION:
In-depth understanding of molecular characteristics of gastric cancer enabled us to realize personalized medicine with targeted agents in gastric cancer treatment.The investigators initiated open-label, randomized, controlled phase II, multi-arm trial comparing targeted therapy based on tumor molecular profiling with standard paclitaxel therapy as second line treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced or metastatic gastric cancer and gastroesophageal junction cancer
2. Eastern Cooperative Oncology Group performance status of 0 to 1
3. Male or female; ≥ 19 years of age
4. On or progression after 1st line palliative chemotherapy
5. Subjects with evaluable lesion (using RECIST 1.1 criteria)
6. Subjects who meet the following criteria:

   * Absolute neutrophil count ≥ 1000 /µL
   * Platelet count ≥ 75,000/ µL
   * Serum creatinine < 1.5 x upper limit of normal or Creatinine clearance ≥60 mL/min
   * aspartate aminotransferase and alanine transaminase 3 x upper limit of normal

Exclusion Criteria:

* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2024-03 (Actual)

PRIMARY OUTCOMES:
progression free survival | 6 weeks
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young Rha, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Yonsei University Health System, Yonsei Cancer Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee CK, Kim HS, Jung M, Kim H, Bae WK, Koo DH, Jeung HC, Park SR, Hwang IG, Zang DY, Lee HW, Park S, Nam CM, Chung HC, Rha SY. Open-Label, Multicenter, Randomized, Biomarker-Integrated Umbrella Trial for Second-Line Treatment of Advanced Gastric Cancer: K-Umbrella Gastric Cancer Study. J Clin Oncol. 2024 Jan 20;42(3):348-357. doi: 10.1200/JCO.23.00971. Epub 2023 Oct 26. PMID 37883723